CLINICAL TRIAL: NCT00589589
Title: Computer Decision Support to Achieve Glycemic Control in the ICU
Acronym: EndoTool
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: United States Army Institute of Surgical Research (U.S. Federal Agency)
Responsible Party: Principal Investigator, Elizabeth Mann, Administrator, United States Army Institute of Surgical Research
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: H-07-040
Record Dates: First submitted 2007-12-24; First posted 2008-01-09 (Estimated); Last update posted 2015-09-03 (Estimated); Status verified 2015-09

CONDITIONS: Burns; Hypoglycemia
Keywords: burns; hypoglycemia; hyperglycemia; glucose monitoring
MeSH Terms: conditions — Burns; Hypoglycemia; Hyperglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Active Comparator)
  Interventions: Device: Endo Tool

INTERVENTIONS:
Device: Endo Tool — Computer tool to help achieve glucose control
  Other Names: Computer Software for glucose control

SUMMARY:
This study is intended to fill the knowledge gap regarding the burn population with research that achieves scientific merit. we will determine the effectiveness of the computer decision support system (CDSS) to facilitate glucose management in the critically ill burn patient.

The EndoTool™ computer decision support system will achieve glycemic control (defined as 80-110 mg/dL) in a shorter time, reduce glycemic excursion outside of target range, and reduce incidence of hypoglycemia (blood glucose less than 50 mg/dL) in the critically ill burn patient compared to the standard of care USAISR insulin titration protocol (Appendix A).

DETAILED DESCRIPTION:
This is a prospective, paired, randomized, cross-over design, with two groups: current standard of care using the USAISR Burn Center insulin titration nomogram (Appendix A) and insulin management using EndoTool™ (MD Scientific, LLC) decision support software. Patients will thus serve as their own controls.

Upon admission to the burn ICU, patients expected to require continuous insulin infusion for a minimum of 7 days will be placed on EndoTool™ CDSS for the first 24 hours of glycemic management. At the 24 hour mark the patients will be randomly assigned to either the CDSS or standard of care group in pairs. Thus, the first subject will be randomized to a group and the second subject will be placed in the alternate group. This method will ensure equal numbers of patients are enrolled in each group to eliminate bias of timing of intervention due to the effect of increasing insulin resistance over time demonstrated in the burn population (Pidcoke, unpublished, USAISR).

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* military or civilian burns on continuous insulin infusion for 7 days

Exclusion Criteria:

* not expected to receive insulin for 7 days
* less than 18 years old
* enrolled in the Continuous Glucose monitoring Study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-01; Primary Completion 2010-09 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Time spent in target glucose range of 80-110 mg/dL. | 48 hours

SECONDARY OUTCOMES:
Time to achieve target glucose of 80-110 mg/dL and number of hypoglycemic events less than 80 and 50 mg/dL. | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A Mann, RN, MSN, Principal Investigator — United States Army Institute of Surgical Research
Locations (1):
- US Army Institute of Surgical Research, Fort Sam Houston, Texas, United States

REFERENCES:
- [Background] Van den Berghe G, Wouters PJ, Bouillon R, Weekers F, Verwaest C, Schetz M, Vlasselaers D, Ferdinande P, Lauwers P. Outcome benefit of intensive insulin therapy in the critically ill: Insulin dose versus glycemic control. Crit Care Med. 2003 Feb;31(2):359-66. doi: 10.1097/01.CCM.0000045568.12881.10. PMID 12576937